CLINICAL TRIAL: NCT05109026
Title: Connect-5 Needs Assessment to Identify Requirements of a Rural Irish Community Related to a an Online Digital Platform Solution, Designed to Change Behaviour, Related to Lifestyle Medicine and Mental Health.
Brief Title: Connect-5 Needs Assessment Survey to Identify Healthy Lifestyle Requirements of a Rural Irish Community
Acronym: CONNECT-5
Status: Completed | Type: Observational
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Private Philanthropic Funder (Other)
Responsible Party: Principal Investigator, Padraic Dunne, Principal Investigator, Royal College of Surgeons, Ireland
Other Study IDs: Connect-5 Needs Assessment
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Healthy Lifestyle
Keywords: Survey; Interviews; Needs Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Older people: Members of the population aged 65 years and older.
- Recent migrants: Members of the population who are recent migrants to the community.
- Members of the travelling community: Members of the population who are members of the travelling community.
- Perinatal women.: Members of the population who are pregnant or within a year of giving birth.
- Lone-parents: Members of the population who are raising children alone.
- Individuals with physical disabilities: Members of the population who have a physical disability.
- Secondary school students: Members of the population attending secondary school.
- Remote workers: Members of the population currently working from home.

SUMMARY:
This is an anonymous needs assessment survey of the population of an Irish urban town. We plan to collect anonymous survey data in order to better understand residents needs and to determine the desired functionality of a new coach-led wellness app operated by our partners. This platform is currently trialled for health care professionals working in the RCSI Hospital Group. The survey will collect information on participants demographics, their lifestyle (including sleep, exercise, food, relationships, meaning and purpose, substance use and stress management). We will also ask participants about their use of wellness apps to support healthy choices related to their lifestyle. We also plan to conduct a qualitative assessment to further explore needs related to lifestyle health in specific cohorts, namely, older people (65 years and older), recent migrants, members of the travelling community, perinatal women, lone-parents, individuals with physical disabilities, secondary school students and remote workers.

DETAILED DESCRIPTION:
There has been an increase in lifestyle related diseases worldwide. Living a healthy lifestyle is important to prevent lifestyle-related diseases such as heart disease, obesity, diabetes, mental health issues, certain cancers, autoimmunity and gastro-intestinal disease. The economic impact of these lifestyle-related diseases in Europe alone is set to exceed €200 billion by 2030. Worldwide, one in five people are at an increased risk of developing severe COVID-19, mostly as a result of underlying lifestyle-related diseases. Additionally, global efforts to manage COVID-19 infection have disrupted regular care required by those with these issues. Dealing with this requires that people better manage their own health and address lifestyle related factors that increase the risk associated with such diseases, including inactivity, substance abuse and unhealthy diet. These risk factors are modifiable and can be reduced by health interventions and tools to support a healthy lifestyle.

The COVID-19 pandemic caused prolonged feelings of fear, uncertainty and isolation among the general population. This is likely to impact vulnerable members of society, such as young people, elderly people and those in ethnic minority communities in greater proportions. Children and adolescents are experiencing increased adverse mental health effects such as social isolation, loneliness, depression and anxiety, during the Covid-19 pandemic. Irish adults aged 70 and over have reported worse mental health and increased feelings of loneliness due to cocooning throughout the pandemic. This social isolation and loneliness puts them at increased risk of cognitive and cardiovascular decline. It is important that we prioritise the development of strategies to maintain social engagement, manage loneliness and encourage continued physical activity among older people.

Work habits are currently changing at a rapid pace. Significant sections of our workforces are now working from home and at least 50% are expected to remain at home, even after the current pandemic has resolved. Reports indicate that a significant proportion of this workforce is experiencing issues with disconnection and mental health. As a result, understanding the impact of remote and flexible working arrangements on employee health and mental wellbeing has been included as a research priority within psychological science. While there is evidence that remote working has positive effects on well-being, these effects are not consistent. Remote working may also lead to greater levels of professional isolation, reduced work-life balance, increase work-related fatigue and have negative impacts on well-being. This study is being conducted to better understand citizen's needs in relation to living a healthier lifestyle.

ELIGIBILITY:
Inclusion Criteria:

- Participants will be members of the urban town being studied.

Exclusion Criteria:

- Non a member of the urban town being studied.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We aim to collect survey data from at least 1,820 participants (20% response rate).
  We will conduct interviews with up to 5 members of each target cohort from the community ( older people, recent migrants, members of the travelling community, perinatal women, lone-parents, individuals with physical disabilities, and remote workers).
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Needs assessment survey | January 2022-February 2022
  An anonymous needs assessment survey (online and hard copies) will be conducted.
Needs assessment interivews | January 2022-March 2022
  Anonymous qualitative interviews will be conducted in conjunction with community liaison officers, over the telephone with up to 5 members of the following target groups - older people (65 years and older), recent migrants, members of the travelling community, perinatal women, lone-parents, individuals with physical disabilities, and remote workers.
Analysis | March 2022- April 2022
  Analysis of summary anonymous aggregate data will be used to inform future stages of this research.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Positive Healthy Sciences, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
Only summary aggregate data will be shared.

REFERENCES:
- [Background] Ng R, Sutradhar R, Yao Z, Wodchis WP, Rosella LC. Smoking, drinking, diet and physical activity-modifiable lifestyle risk factors and their associations with age to first chronic disease. Int J Epidemiol. 2020 Feb 1;49(1):113-130. doi: 10.1093/ije/dyz078. PMID 31329872
- [Background] Hyland P, Shevlin M, McBride O, Murphy J, Karatzias T, Bentall RP, Martinez A, Vallieres F. Anxiety and depression in the Republic of Ireland during the COVID-19 pandemic. Acta Psychiatr Scand. 2020 Sep;142(3):249-256. doi: 10.1111/acps.13219. Epub 2020 Aug 9. PMID 32716520
- [Background] Nearchou F, Flinn C, Niland R, Subramaniam SS, Hennessy E. Exploring the Impact of COVID-19 on Mental Health Outcomes in Children and Adolescents: A Systematic Review. Int J Environ Res Public Health. 2020 Nov 16;17(22):8479. doi: 10.3390/ijerph17228479. PMID 33207689
- [Background] Loades ME, Chatburn E, Higson-Sweeney N, Reynolds S, Shafran R, Brigden A, Linney C, McManus MN, Borwick C, Crawley E. Rapid Systematic Review: The Impact of Social Isolation and Loneliness on the Mental Health of Children and Adolescents in the Context of COVID-19. J Am Acad Child Adolesc Psychiatry. 2020 Nov;59(11):1218-1239.e3. doi: 10.1016/j.jaac.2020.05.009. Epub 2020 Jun 3. PMID 32504808
- [Background] Bailey T, Hastings RP, Totsika V. COVID-19 impact on psychological outcomes of parents, siblings and children with intellectual disability: longitudinal before and during lockdown design. J Intellect Disabil Res. 2021 May;65(5):397-404. doi: 10.1111/jir.12818. Epub 2021 Feb 25. PMID 33634520
- [Background] Ward MP. SARS-CoV-2, where to now? Transbound Emerg Dis. 2020 Jul;67(4):1411-1413. doi: 10.1111/tbed.13654. Epub 2020 Jun 19. No abstract available. PMID 32562349
- [Background] Fried L, Prohaska T, Burholt V, Burns A, Golden J, Hawkley L, Lawlor B, Leavey G, Lubben J, O'Sullivan R, Perissinotto C, van Tilburg T, Tully M, Victor C. A unified approach to loneliness. Lancet. 2020 Jan 11;395(10218):114. doi: 10.1016/S0140-6736(19)32533-4. No abstract available. PMID 31929010
- [Background] Valtorta NK, Kanaan M, Gilbody S, Ronzi S, Hanratty B. Loneliness and social isolation as risk factors for coronary heart disease and stroke: systematic review and meta-analysis of longitudinal observational studies. Heart. 2016 Jul 1;102(13):1009-16. doi: 10.1136/heartjnl-2015-308790. Epub 2016 Apr 18. PMID 27091846
- [Background] O'Connor DB, Aggleton JP, Chakrabarti B, Cooper CL, Creswell C, Dunsmuir S, Fiske ST, Gathercole S, Gough B, Ireland JL, Jones MV, Jowett A, Kagan C, Karanika-Murray M, Kaye LK, Kumari V, Lewandowsky S, Lightman S, Malpass D, Meins E, Morgan BP, Morrison Coulthard LJ, Reicher SD, Schacter DL, Sherman SM, Simms V, Williams A, Wykes T, Armitage CJ. Research priorities for the COVID-19 pandemic and beyond: A call to action for psychological science. Br J Psychol. 2020 Nov;111(4):603-629. doi: 10.1111/bjop.12468. Epub 2020 Jul 19. PMID 32683689